CLINICAL TRIAL: NCT00361244
Title: A Phase I/II Study of SU011248 (Sutent) in Combination With Irinotecan and Cetuximab as a Second Line Regimen for Patients With Stage IV Colorectal Cancer
Brief Title: SU011248 in Combination With Irinotecan and Cetuximab as a Second Line Regimen for Stage IV Colorectal Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Slow Accrual
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Beth Israel Deaconess Medical Center (Other); Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Andrew X. Zhu, MD, Physician Hematology/Oncology, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 05-439
Record Dates: First submitted 2006-08-04; First posted 2006-08-08 (Estimated); Last update posted 2017-02-17 (Actual); Status verified 2017-02

CONDITIONS: Colorectal Carcinoma
Keywords: Sutent
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Sunitinib; Irinotecan; Cetuximab

INTERVENTIONS:
Drug: SU011248 — Given orally in the morning for two weeks followed by a one week rest period (one cycle equals 21 days). Participants may continue to receive study treatment as long as their disease does not progress and they do not experience any serious side effects.
Drug: Irinotecan — Given intravenously on days 1 and 8 of each 21-day cycle. Participants may continue to receive study treatment as long as their disease does not progress and they do not experience any serious side effects.
Drug: Cetuximab — Given intravenously on days 8 and 15 of each 21-day cycle. Participants may continue to receive study treatment as long as their disease does not progress and they do not experience any serious side effects.

SUMMARY:
The purpose of this study is to determine the safety of SU011248 and the highest dose of this drug that can be given safely in combination with the chemotherapy drugs irinotecan and cetuximab. Laboratory studies have shown that SU011248 may block the growth of blood vessels in tumors, which may prevent tumors from growing any further. Other studies have demonstrated the possibility that SU011248 may enhance the anti-tumor activity of other chemotherapy drugs such as irinotecan and cetuximab.

DETAILED DESCRIPTION:
* Participants will be given a supply of SU011248 capsules to take at home in the morning for two weeks. After taking the capsules for two weeks, there will be a one-week rest period.
* Irinotecan will be administered on days 1 and 8 of every 21-day cycle as an intravenous infusion over 90 minutes. Cetuximab will be administered intravenously on days 1, 8 and 15 of every 21-day cycle. The first treatment of cetuximab is a larger dose. Beginning with the second treatment, the participant will receive a smaller dose of cetuximab.
* Blood work will be repeated at every clinic visit on days 1 and 8. During cycle 1, blood will also be drawn on day 15.
* Tumor assessments will be repeated after 6 weeks, 12 weeks, and every 9 weeks thereafter, and will be assessed by both a CT scan of the abdomen, pelvis, and a chest x-ray. MUGA scans will be repeated every 4 cycles (12 weeks).
* Participants may continue to receive cycles of study treatment as long as their disease does not progress and they do not experience any serious side effects.

ELIGIBILITY:
Inclusion Criteria:

* Histologic proof of adenocarcinoma of the colon or rectum with evidence of metastatic disease. The site of the primary lesion must be or have been confirmed endoscopically, radiologically, or surgically to be or have been in the large bowel
* Patients must have received one (and only one) prior chemotherapy regimen for metastatic disease using 5-FU/LV or Xeloda in combination with oxaliplatin and Avastin.
* > 4 weeks must have elapsed from the time of major surgery
* > 2 weeks must have elapsed from the time of minor surgery
* > 4 weeks must have elapsed from the time of major radiotherapy
* Normal organ and marrow function
* Measurable disease be RECIST criteria
* Older than 18 years of age
* ECOG performance status of 0-1
* Life expectancy > 12 weeks

Exclusion Criteria:

* Previous treatment with irinotecan, cetuximab or SU011248
* Any of the following within the 12 months prior to study drug administration: severe/unstable angina; myocardial infarction; symptomatic congestive heart failure; cerebrovascular accident; or transient ischemic attack.
* Known brain metastases or carcinomatous meningitis
* Uncontrolled serious medical or psychiatric illness
* NCI CTCAE grade 3 or greater hemorrhage within 4 weeks of starting study treatment
* Uncontrolled hypertension
* Diagnosis of any secondary malignancies with the last 5 years, except for adequately treated basal cell carcinoma, squamous cell skin cancer, localized prostate cancer with a normal PSA within the past 3 months, in situ bladder cancer, or in situ cervical cancer
* Pregnant or breastfeeding
* Concurrent treatment on another clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2006-07 (Actual); Primary Completion 2007-10 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
To determine the maximum tolerated dose of SU011248 when given in combination with irinotecan and cetuximab in patients with previously treated locally advanced, locally recurrent, or metastatic colorectal adenocarcinoma | 1 year
To determine the response rate of SU011248 when given in combination with irinotecan and cetuximab in this patient population.

SECONDARY OUTCOMES:
To evaluate the toxicities of this combination of drugs in this patient population | 1 year
to assess overall survival, progression-free survival, time to progression and duration of response.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew X. Zhu, MD, Principal Investigator — Massachusetts General Hospital
Locations (3):
- United States (3):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts